CLINICAL TRIAL: NCT00040911
Title: A Randomized Study Of Electroacupuncture Treatment For Delayed Chemotherapy-Induced Nausea And Vomiting In Patients With Pediatric Solid Tumors
Brief Title: Electroacupuncture in Treating Delayed Nausea and Vomiting in Patients Receiving Chemotherapy For Newly Diagnosed Childhood Sarcoma, Neuroblastoma, Nasopharyngeal Cancer, Germ Cell Tumors, or Hodgkin Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ACCL04C2; NCCAM-02-AT-0172; NCI-02-AT-0172 (Other: NCI); COG-ACCL04C2 (Other: Children's Oncology Group); CDR0000069419 (Other: Clinical Trials.gov); NCT00034411 (obsolete NCT alias); NCT00034996 (obsolete NCT alias)
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Brain Tumors; Central Nervous System Tumors; Childhood Germ Cell Tumor; Extragonadal Germ Cell Tumor; Head and Neck Cancer; Lymphoma; Nausea; Vomiting; Neuroblastoma; Ovarian Cancer; Sarcoma
Keywords: nausea and vomiting; localized osteosarcoma; metastatic osteosarcoma; nonmetastatic childhood soft tissue sarcoma; metastatic childhood soft tissue sarcoma; previously untreated childhood rhabdomyosarcoma; localized Ewing sarcoma/peripheral primitive neuroectodermal tumor; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; childhood teratoma; childhood extragonadal germ cell tumor; childhood malignant testicular germ cell tumor; childhood malignant ovarian germ cell tumor; childhood central nervous system germ cell tumor; localized resectable neuroblastoma; localized unresectable neuroblastoma; disseminated neuroblastoma; regional neuroblastoma; stage 4S neuroblastoma; stage I lymphoepithelioma of the nasopharynx; stage I squamous cell carcinoma of the nasopharynx; stage II lymphoepithelioma of the nasopharynx; stage II squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage I adult Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage II childhood Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms; Head and Neck Neoplasms; Lymphoma; Nausea; Vomiting; Neuroblastoma; Ovarian Neoplasms; Sarcoma; Osteosarcoma; Neuroectodermal Tumors, Primitive, Peripheral; Teratoma; Testicular Neoplasms; Ovarian Germ Cell Cancer; Hodgkin Disease | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (alternative medicine procedure) (Experimental): Patients undergo electroacupuncture therapy to specific acupuncture points on the arms and legs over 25 minutes twice daily on days 1 and 2 and then once daily on days 3-7 during week 1 of chemotherapy course 1 (9 acupuncture treatments total).
  Interventions: Procedure: electroacupuncture therapy; Procedure: quality-of-life assessment
- Arm II (alternative medicine procedure) (Sham Comparator): Patients undergo electroacupuncture therapy to sham points on the arms and legs as in arm I.
  Interventions: Procedure: sham intervention; Procedure: quality-of-life assessment

INTERVENTIONS:
Procedure: electroacupuncture therapy
  Arms: Arm I (alternative medicine procedure)
Procedure: sham intervention — Undergo electroacupuncture therapy to sham points
  Arms: Arm II (alternative medicine procedure)
Procedure: quality-of-life assessment — Ancillary studies

SUMMARY:
RATIONALE: Electroacupuncture may help to reduce or prevent delayed nausea and vomiting in patients treated with chemotherapy.

PURPOSE: This randomized clinical trial is studying the effectiveness of electroacupuncture in treating delayed nausea and vomiting in patients who are receiving chemotherapy for newly diagnosed childhood sarcoma, neuroblastoma, nasopharyngeal cancer, germ cell tumors, or Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of electroacupuncture, in terms of reducing acute and delayed chemotherapy-induced nausea, in patients with newly diagnosed pediatric sarcoma, neuroblastoma, nasopharyngeal carcinoma, or germ cell tumors.

Secondary

* Determine the efficacy of this therapy, in terms of reducing delayed chemotherapy-induced emesis, in these patients.
* Determine the efficacy of this therapy, in terms of altering salivary cortisol levels and fasting serum glucose and insulin levels as stress parameters, in these patients.
* Determine the efficacy of this therapy, in terms of improving the quality of life, in these patients.
* Determine the efficacy of this therapy, in terms of reducing acute nausea and emesis, in these patients.

OUTLINE: This is a multicenter, randomized, double-blind study. Patients are stratified according to planned treatment with cisplatin-based chemotherapy (yes vs no) and gender. Patients are randomized to 1 of 2 arms.

* Arm I: Patients undergo electroacupuncture to specific acupuncture points on the arms and legs over 25 minutes twice daily on days 1 and 2 and then once daily on days 3-7 during week 1 of chemotherapy course 1 (9 acupuncture treatments total).
* Arm II: Patients undergo electroacupuncture to sham points on the arms and legs as in arm I.

Quality of life is assessed at baseline, on days 1 and 8 of each treatment course, and then after completion of the study.

PROJECTED ACCRUAL: A total of 65 patients (approximately 32 per arm) will be accrued for this study within 2.5-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed malignancy of 1 of the following types:

  * Pediatric sarcoma
  * Neuroblastoma
  * Nasopharyngeal carcinoma
  * Germ cell tumor
  * Hodgkin lymphoma
* Meets 1 of the following criteria:

  * Eligible for Children's Oncology Group (COG) protocol for sarcoma, neuroblastoma, or germ cell tumor
  * Eligible for NCI Pediatric Oncology Branch (POB) protocol for sarcoma
  * Following COG-approved standard treatment regimen for sarcoma, neuroblastoma, nasopharyngeal carcinoma, or germ cell tumor
  * Enrolled on the POB natural history protocol 98-C-0037
* Planned treatment, according to COG or POB protocols, that includes a cisplatin- and/or doxorubicin-containing regimen for sarcoma, neuroblastoma, nasopharyngeal carcinoma, germ cell tumor, or Hodgkin lymphoma OR either a cyclophosphamide/ifosfamide-doxorubicin-containing or cyclophosphamide/dactinomycin-containing regimen for rhabdomyosarcoma
* No clinical or radiographic signs of spinal cord compression

PATIENT CHARACTERISTICS:

Age:

* 5 to 35

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Platelet count greater than 50,000/mm^3 (transfusion independent)
* No clotting disorders, including hemophilia

Hepatic:

* PT and PTT normal (within 10% of institution's upper limit of normal)

Renal:

* Not specified

Other:

* Not pregnant
* No casting of 1 or more extremities
* No other condition that would preclude access to acupuncture points
* No cognitive impairment

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No prior systemic chemotherapy

Endocrine therapy:

* More than 4 weeks since prior glucocorticoid therapy
* No concurrent glucocorticoid therapy

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No prior acupuncture
* No concurrent anticoagulants

Ages: 5 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2005-04; Primary Completion 2009-10 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Delayed nausea by Marrow Assessment of Nausea and Emesis at 1, 3, and 6 weeks after study completion | 7 days
  A two-sample t-test will be used. In the event the data are not normally distributed in one or both arms, a Wilcoxon rank sum test will be used.

SECONDARY OUTCOMES:
Quality of life by QLQ C-30 at 1, 3, and 6 weeks after study completion | Day 8
Pain by Brief Pain Inventory at 1, 3, and 6 weeks after study completion | Day 1
  It is anticipated that Cochran-Armitage trend tests will be used to compare the results between randomized groups.

CONTACTS AND LOCATIONS:
Overall Officials: Kara Kelly, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States